CLINICAL TRIAL: NCT01579409
Title: " Impact Du Statut Alimentaire Sur La Fonction Vasculaire Avant Et Après Un Petit-déjeuner Standardisé. Une Étude " Exposé/non Exposé " Nichée Dans La Cohorte SUVIMAX2
Brief Title: Impact of Dietary Status on Vascular Function Before and After a Standardized Breakfast. an "exposed/unexposed" Study Embedded in the SUVIMAX2 Cohort
Acronym: Nutri-MicroVas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: C11-20; 2011-A01003-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-04-06; First posted 2012-04-18 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: French PNNS Guidelines in Vascular Function
Keywords: Nutrition; Arterial stiffness; Endothelial dysfunction; Microcirculation; Cardiac autonomic system.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1-25th percentile of the PNNS score (Other)
  Interventions: Other: PNNS guidelines
- 75-100th percentile of the PNNS score (Other)
  Interventions: Other: PNNS guidelines

INTERVENTIONS:
Other: PNNS guidelines — Application of PNNS guidelines

SUMMARY:
In France, primary cardiovascular and metabolic prevention is supported by the French National Program for Nutrition and Health (PNNS: Programme National Nutrition Santé).

The investigators made the hypothesis that, independently of other diseases, the non adherence in PNNS guidelines would lead to arterial stiffness, endothelial dysfunction, change in microcirculation and in cardiac autonomic system. These changes may exist at fasting but also be reinforced after a standardised breakfast.

The investigators aim is to evaluate arterial stiffness, endothelial function, microcirculation and cardiac autonomic system according to PNNS status in a case control study.

DETAILED DESCRIPTION:
This is a case / control pilot nested in SU.VI.MAX 2 (SUpplémentation en VItamines et Minéraux Anti-oXydants) study. The randomized longitudinal placebo controlled SU.VI.MAX study tested the preventive effect of vitamin and antioxidant minerals supplementation on the incidence and the mortality from cardiovascular pathologies and cancers. SU.VI.MAX 2 was the extension of the previous study and included 7200 subjects for whom food habits were known and characterized according to PNNS guidelines (PNNS score).

The subjects will be pre-selected from the original cohort SU.VI.MAX2 if they have a PNNS score in 2007 in the 1-40th or 60-100th percentiles of distribution. If they accept to participate, a new PNNS score will be calculated in 2012-2013 and the subjects in the 1-25th or 75-100th percentiles will be included and explored during one day of participation.

Our aim is to evaluate arterial stiffness, endothelial function, microcirculation and cardiac autonomic system according to PNNS status in a case control study.

Our secondary objective is to evaluate the same parameters in the same subjects but after a breakfast containing 75 g glucose.

ELIGIBILITY:
Inclusion Criteria:

* Social Security affiliation.
* Participation in SU.VI.MAX 2.
* Subjects without legal guardian who can freely agree to participate to the study.
* PNNS score in 2012 lower (cases) or upper (controls) quartile.

Exclusion Criteria:

* Known diabetes or prediabetes before the inclusion.
* History of cardiovascular disease.
* Treatment for hypertension.
* Treatment for dyslipidemia.
* Known Cancer
* Smoking or patients that have stopped smoking less than 3 years
* Cardiac pacemaker

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2014-03-04 (Actual); Study Completion 2014-03-04 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates
  This is a pilot study. Pulse wave velocity, an index of arterial stiffness, was chosen as the primary endpoint. A total of 47 subjects in each group was necessary to detect a difference between groups of 1m/s in pulse wave velocity (standard deviation of 1.7 m/s) with a statistical power of 80%, at fasting.
Peripheral arterial augmentation index (Aix ) | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates
High and low frequency peaks in heart variability spectral analysis | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates
High and low frequency peaks in systolic and diastolic blood pressure spectral analysis | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates
Mean cutaneous blood flow measured by laser doppler flowmetry | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates
Mean cutaneous blood flow measured by laser doppler flowmetry, spectral analysis | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates
Percentage of variation of cutaneous blood flow laser doppler measurements after paced breathing (6/min) | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates
Increase in cutaneous blood flow laser doppler measurements after acetylcholine iontophoresis | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates
Reactive Hyperemia Index after branchial artery occlusion | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates
Aortic , radial,digital artery, systolic, diastolic and pulsatile pressures | During the fasting state, within the hour preceding the standardised breakfast that provides 75 gr of carbohydrates

SECONDARY OUTCOMES:
Comparison of the above mentioned parameters after a standardised breakfast | After the standardised breakfast that provides 75 gr of carbohydrates, hourly for the next 3 hours following the end of the standardised breakfast

CONTACTS AND LOCATIONS:
Overall Officials: Paul Valensi, MD, Study Director — CNRH Ile de france

REFERENCES:
- [Derived] Fysekidis M, Kesse-Guyot E, Valensi P, Arnault N, Galan P, Hercberg S, Cosson E. Association Between Adherence To The French Dietary Guidelines And Lower Resting Heart Rate, Longer Diastole Duration, And Lower Myocardial Oxygen Consumption. The NUTRIVASC Study. Vasc Health Risk Manag. 2019 Oct 30;15:463-475. doi: 10.2147/VHRM.S215795. eCollection 2019. PMID 31802880